CLINICAL TRIAL: NCT05118672
Title: A Multicenter, Randomized, Parallel-group, Double-blind, Comparative Trial of the Superiority of Paracetamol 500mg/Fexofenadine 60mg/Phenylephrine 20mg Fixed-dose Combination Versus Placebo in the Symptomatic Treatment of Flu and Cold
Brief Title: Phase 3 Clinical Trial to Evaluate Paracetamol /Fexofenadine /Phenylephrine in Flu and Cold Treatment
Acronym: RESFRIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EF175
Record Dates: First submitted 2021-10-05; First posted 2021-11-12 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-03

CONDITIONS: Cold; Flu Symptom
MeSH Terms: conditions — Common Cold | interventions — Drugs, Investigational; Acetaminophen; fexofenadine; Phenylephrine

STUDY DESIGN:
Intervention Model Description: Adult participants (aged ≥ 18 years) of both sexes with common cold or flu will be randomized in a 1:1 ratio to receive the experimental drug (paracetamol 500 mg / fexofenadine 60 mg / phenylephrine 20 mg) or placebo, in the dosage of one (01) film-coated tablet every eight (08) hours, for 3 to 7 days.
  Randomized participants will be instructed to use the study treatment uninterruptedly, every eight (08) hours, for three (03) days, and may, after that, discontinue treatment at any time if they experience no more symptoms.
Who Masked: Participant, Investigator
Masking Description: Group 1: Eurofarma Laboratórios SA paracetamol 500mg / fexofenadine 60mg / phenylephrine 20mg FDC (experimental drug).
  Group 2: Placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental drug (paracetamol 500mg / fexofenadine 60mg / phenylephrine 20mg) (Experimental): Group 1: paracetamol 500mg / fexofenadine 60mg / phenylephrine 20mg FDC (experimental drug).
  Interventions: Drug: Experimental drug (paracetamol 500mg / fexofenadine 60mg / phenylephrine 20mg)
- Placebo group (Placebo Comparator): Group 2: Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Experimental drug (paracetamol 500mg / fexofenadine 60mg / phenylephrine 20mg) — Subjects randomized to this group will receive one (01) experimental drug film-coated tablet every eight (08) hours for three (03) days (nine [09] dosage administration). Subjects will be instructed to, thereafter, maintain treatment at the same dosage (one [01] film-coated tablet every eight [08] hours) in case of persistence of symptoms, discontinuing treatment when they present with no symptoms.
  Other Names: EF175
  Arms: Experimental drug (paracetamol 500mg / fexofenadine 60mg / phenylephrine 20mg)
Drug: Placebo — Subjects randomized to this group will receive one (01) experimental drug film-coated tablet every eight (08) hours for three (03) days (nine [09] dosage administration). Subjects will be instructed to, thereafter, maintain treatment at the same dosage (one [01] film-coated tablet every eight [08] hours) in case of persistence of symptoms, discontinuing treatment when they present with no symptoms.
  Other Names: EF175 Placebo
  Arms: Placebo group

SUMMARY:
A Phase 3, multicenter, Randomized, Double-blind, comparative clinical trial to evaluate the association of paracetamol 500mg + Fexofenadine 60mg + Phenylephrine 20mg in the flu and common cold treatment.

⚠️Study will only be conducted in research centers in Brazil (please do not send e-mail if your center is outside brazil).

DETAILED DESCRIPTION:
A multicenter, randomized, double-blind, parallel-group, superiority, placebo control clinical trial.

Adult patients (aged ≥ 18 years) of both sexes with common cold or flu will be randomized in a 1:1 ratio to receive the experimental drug (paracetamol 500mg / fexofenadine 60mg / phenylephrine 20mg) or placebo, in the dosage of one (01) film-coated tablet every eight (08) hours, for 3 to 7 days.

The primary superiority assessment will be carry out compared the experimental drug to placebo in the relief of cold and flu symptoms through the absolute variation of the overall score obtained in the symptom assessment questionnaire after treatment start.

⚠️Study will only be conducted in research centers in Brazil (please do not send e-mail if your center is outside brazil).

ELIGIBILITY:
Inclusion Criteria:

* Common cold: presence of moderate to severe nasal congestion AND moderate to severe runny nose AND at least one (01) of the following moderate to severe symptoms: sneezing, headache, myalgia, sore throat, throat pain, dysphonia, cough and fever.

Duration of symptoms ≤ 48 hours at screening. Informed Consent Form (ICF) signed before carrying out any study procedure.

Exclusion Criteria:

* Presence of significant septum deviation, compatible with impaired nasal ventilatory function, at the investigator's discretion.
* Presence of nasal polyposis to previous rhinoscopy.
* Known hypersensitivity to any component of the experimental drug formulation.
* Required antibiotic therapy for upper airway infection treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 567 (Actual)
Dates: Start 2025-03-26 (Actual); Primary Completion 2025-08-26 (Actual); Study Completion 2025-08-26 (Actual)

PRIMARY OUTCOMES:
Relief of cold and flu symptoms | 26 hours
  absolute variation of the overall score obtained in the symptom assessment questionnaire (Likert Scale), in which nasal congestion, runny nose, sneezing, headache, myalgia, sore throat, throat pain hoarseness, cough and fever will be assessed on a 4-point categorical scale (0 = absent, 1 = mild, 2 = moderate and 3 = severe) after administration of the first dose of the study treatment from baseline.
  The overall symptom score will be determined by the sum of the points assigned to the individual symptoms. The baseline overall score will vary in the interval of 6 to 30 points, ranging from 0 to 30 points in the other assessments, and the higher the score, the worse the subject's symptoms

SECONDARY OUTCOMES:
overall efficacy of the experimental drug | 11 days
  subject's treatment overall evaluation 3 (±1) days after the administration of the first dose of study treatment from baseline.
efficacy of the experimental drug on the nasal congestion symptoms | 3 hours (± 30 minutes), 26 (± 2) hours and 3 (± 1) days after administration
  Proportion of subjects with improved nasal congestion and runny nose 3 hours (± 30 minutes), 26 (± 2) hours and 3 (± 1) days after administration of the first dose of the study treatment from baseline, being considered improvement the reduction of at least one point on the 4-point categorical Likert scale (0 = absent, 1 = mild, 2 = moderate, and 3 = severe).
duration of the experimental drug treatment | 7 days
  Duration (in days) of study treatment
use of rescue medication | 7 days
  Amount (in number of tablets) of rescue medication used.

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Eurofarma Laboratórios S.A, São Paulo, São Paulo
  - Clinica de Alergia Martti Antila, Sorocaba, São Paulo

IPD SHARING:
Plan to Share IPD: No